CLINICAL TRIAL: NCT02997826
Title: Effect of Infant Formula Consumption on Infant Growth From 0 to 6 Months
Brief Title: Effect of Infant Formula Intake on Infant Growth From 0 to 6 Months.
Acronym: BABYMILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Professor, Institut Pasteur de Lille
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A01403-48
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Child Development

ARMS (1):
- 1 to 21-days old child (Other)
  Interventions: Other: Infantil formula

INTERVENTIONS:
Other: Infantil formula

SUMMARY:
From birth to 5 months, milk is the essential and unique food of the newborn. The French National Nutrition Program (PNNS) recommends exclusive breastfeeding "up to 6 months and at least 4 months for a healthy benefit". However, only 36% of infants 0-6 months of age are exclusively breastfed worldwide. Some mothers choose to give infant formula to their baby in the first few months of life. This decision may be a personal choice or be imposed by pathophysiological situations.

The nutritional requirements of the infant are specific, which implies adequate nutrition. Infant formulas and follow-up formulas are therefore complex products, specially developed for a group of vulnerable consumers. In fact, the compositional and information requirements for infant formula are highly regulated.

Even clinical studies are not required to market an infant formula, it is important to obtain objective date on infant growth. Therefore, this study proposes to evaluate the effect of the consumption of an infant formula on the growth of infants from 0 to 6 months in comparison with the growth curves of the World Health Organization (WHO).

ELIGIBILITY:
Inclusion Criteria:

* 0 to 3 weeks
* Infants whose mothers do not wish or can not breastfeed for personal or medical reasons
* Child followed by a general practitioner or pediatrician
* Informed consent form signed by the legal representatives of the subject
* Commitment of legal representatives to follow the constraints generated by the study
* Insured

Exclusion Criteria:

* Nursing mother
* Infant born prematurely before 37 weeks of amenorrhea
* Child allergic to cow's milk proteins
* Pathological pregnancy (hypertension, infection, gestational diabetes, etc.);
* Chronic or acute illness (metabolic or neuromuscular diseases, epilepsy, asthma, diabetes, digestive, renal, cardiac or haematological diseases);
* Incapacity for the legal representative(s) to understand or adhere to the protocol
* Mother smoking or vapoting during pregnancy;
* Subject involved in another clinical study or in an exclusion period from another study
* Legal representatives deprived of liberty
* Legal representatives in a position to judicial protection
* Weight of the subject according to age and sex, not included between the 3rd and the 97th percentile of the WHO Child Growth Standards
* Subject height according to age and sex, not between the 3rd and the 97th percentile of the WHO Child Growth Standards
* BMI of the subject according to age and sex, not included between the 3rd and the 97th percentile of the WHO Child Growth Standards
* Head circumference of the subject according to age and sex, not included between the 3rd and the 97th percentile of the WHO Child Growth Standards

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Weight evolution of infants fed with infant formula | from 0 to 3 months

SECONDARY OUTCOMES:
Weight evolution of infants fed with infant formula | from 0 to 6 months
Height evolution of infants fed with infant formula | from 0 to 6 months
Head circumference evolution of infants fed with infant formula | from 0 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- Institut Pasteur de Lille, Lille, France